CLINICAL TRIAL: NCT02114762
Title: Balloon Dilation in Selected Subjects With Refractory Eustachian Tube Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Cuneyt M. Alper, Professor of Otolaryngology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO13120437; R21DC013167 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Eustachian Tube Dysfunction
Keywords: otitis media; eustachian tube; eustachian tube dysfunction; eustachian tube function testing
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon dilation of the Eustachian tube (Experimental): Insertion and inflation of balloon into Eustachian tube for up to 1 minute
  Interventions: Procedure: Balloon dilation of the Eustachian tube

INTERVENTIONS:
Procedure: Balloon dilation of the Eustachian tube — Insert a balloon into one Eaustachian tube and inflate it for up to one minute. The balloon is then removed.
  Other Names: Balloon tuboplasty

SUMMARY:
This study evaluates the usefulness and safety of using a balloon to dilate (make larger) the Eustachian tube in adults who have middle-ear disease due to Eustachian tube dysfunction.

DETAILED DESCRIPTION:
The Eustachian tube is a biological tube that connects the back of the nose to the middle ear. It is usually closed but needs to be actively opened by the action of certain muscles during swallowing, yawning, and other activities which keeps the air pressure in the middle ear (the part of the ear behind the eardrum) the same as the air pressure in the environment. If the Eustachian tube does not open during swallowing, the middle-ear pressure progressively decreases and persons may have the feeling of a "stuffed up" and/or "full" middle ear, may have difficulty hearing and/or may develop fluid in their middle ear.

The usual treatment for a Eustachian tube that does not open well is to insert a tiny tube (called a ventilation or tympanostomy tube) into the eardrum to keep the air pressure in the middle ear the same as in the environment. However, those tubes naturally "fall out" over time, and if the Eustachian tube opening function had not improved while they were in place, new tubes will need to be inserted. In the past few years, doctors in the U.S. and Europe described a simple procedure called "balloon dilation of the Eustachian tube" (BDET) or "balloon tuboplasty" that they believe corrects the underlying cause of Eustachian tube dysfunction and resolves its symptoms, signs and consequences. For that procedure, a tiny balloon is inserted into the Eustachian tube, inflated to physically open the Eustachian tube, deflated and then removed. Doctors who have used the method in adults and children with symptoms of Eustachian tube dysfunction reported that BDET is safe and causes a short-term and, perhaps, a long-term resolution of symptoms. However, no one has measured Eustachian tube function before and after the procedure, and it is not known if BDET truly improves that function or not, and if so, how that function is changed.

In this study, we will enroll adult subjects with a tympanostomy tube inserted into at least one eardrum or a chronic perforation in at least one eardrum for physician-diagnosed Eustachian tube dysfunction or middle-ear fluid and document the presence/absence of measurable Eustachian tube dysfunction using standard tests. If present, we will determine if the Eustachian tube dysfunction improves after medical treatment of other diseases known to cause Eustachian tube dysfunction. If the Eustachian tube dysfunction does not significantly improve, we will perform the BDET procedure and measure the change in Eustachian tube function at different times after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* has functional ventilation tube or a chronic perforation in at least one ear;
* history of Eustachian tube dysfunction and/or otitis media with effusion;
* history of middle-ear effusion at least once;
* otherwise healthy except for possible gastro-esophageal reflux disease (GERD), allergies, sinusitis;
* BMI of less than 35;
* no history of difficult intubation;
* no known family history of malignant hyperthermia.

Exclusion Criteria:

* history of adverse reaction to any study-related medication and a suitable alternative is not available;
* current or past history of cancer;
* current or past history of vestibular pathology or cranial base surgery;
* craniofacial dysmorphology (examples: down syndrome, cleft palate);
* pregnancy or "at risk" and not using contraception;
* patulous Eustachian tube;
* non-patent nasal cavity;
* adenoids that block the Eustachian tube orifice;
* blood pressure greater than 140/90;
* had experimental drug or procedure in the previous 3 months;
* allergic to eggs, egg products, soy, or soy products;
* previously underwent balloon dilation of the Eustachian tube.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Eustachian tube function testing | 1 month post-operatively
  opening pressure, closing pressure, passive resistance

SECONDARY OUTCOMES:
Eustachian tube function testing | 3 months post-operatively
  opening pressure, closing pressure, passive resistance
Eustachian tube function testing | 6 months post-operatively
  opening pressure, closing pressure, passive resistance
Eustachian tube function testing | 4 weeks after beginning medical treatment
  opening pressure, closing pressure, passive resistance

OTHER OUTCOMES:
video-endoscopy | entry visit
  ability of video-endoscopy to diagnose anatomic cause of eustachian tube dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607